CLINICAL TRIAL: NCT00411164
Title: A Phase 3, Randomized, Double-Blind, Fixed-Dose, Parallel Group Comparison of Controlled-Release Hydromorphone HCI vs Placebo in Subjects With Osteoarthritis
Brief Title: A Study to Evaluate the Effectiveness and Safety of Slow Release Hydromorphone HCL for Treatment of Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013273
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: knee pain; hip pain; opioid
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

INTERVENTIONS:
Drug: OROS hydromorphone HCI (slow release)

SUMMARY:
The purpose of this study was to compare the analgesic (a drug that relieves pain) effectiveness and safety of OROS hydromorphone HCI (slow release) 8 mg and 16 mg to placebo (no drug) in patients with osteoarthritis (OA).

DETAILED DESCRIPTION:
This was a phase 3, randomized (patients are assigned different treatments based on chance), placebo-controlled, double-blind, fixed-dose, parallel-group, multicenter study in adult patients with OA (osteoarthritis) who were unable to consistently control or treat their pain with nonopioid medications, or who had received an opioid for treatment of pain. Eligible patients were randomized in an equal ratio to receive 1 of 3 treatments: OROS hydromorphone HCI (slow release) 8mg, OROS hydromorphone HCI (slow release) 16 mg, or placebo (no drug). All patients could take acetaminophen (less than or equal to 2000 mg per day) as rescue medication for osteoarthritic pain. Rescue medication was not permitted during the washout period or 6 hours before an assessment of effectiveness. The study was comprised of the following periods: an analgesic (pain reliever) taper and washout period (less than or equal to 2 weeks), a Titration (increase)Phase (less than or equal to 16 days), a Maintenance Phase (12 weeks), and a study drug taper period (less than or equal to 1 week). At the end of the washout period, all patients received OROS hydromorphone HCI (slow release) 8 mg or matching placebo to be taken once daily. After 1 week, patients were to return to the study site and receive new supplies of study drug. During the second week of titration (increase), patients randomized to the OROS hydromorphone (slow release) 16 mg group had their dose increased from 8 mg daily to 16 mg daily of OROS hydromorphone (slow release). No dose adjustments were allowed. After completing the Maintenance Phase or upon early termination, study drug was tapered for up to 1 week as follows: one 8 mg tablet or placebo once daily for the first 2 days then taken every other day as appropriate to taper off the study medication. Safety assessments of physical examination, vital signs, labs and adverse event reporting were done at baseline, termination throughout the study. The primary measurement was the time-interval weighted area under the curve(AUC) divided by the maximum AUC benefit possible for an individual. The AUC was a measure of cumulative pain intensity differences from baseline for the Titration and Maintenance phases. At termination, patients were assigned their baseline pain value for the remainder of the trial, baseline observation carried forward (BOCF) or the last available pain value for the remainder of the trial, last observation carried forward (LOCF). Western Ontario and McMaster Osteoarthritis Index (WOMAC) overall index score, physical function, joint stiffness subscales were analyzed using the AUC ratio and change from baseline using no imputation, and the baseline observation carried forward (BOCF) and last observation carried forward (LOCF) imputation methods. The medical outcome study (MOS) sleep scale was also analyzed per protocol. OROS hydromorphone (slow release) 8 mg and 16 mg tablets and placebo taken orally once daily for 17 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a negative pregnancy test at screening and be postmenopausal for at least 1 year or surgically sterile or practicing a medically recognized contraceptive program
* Patient has been diagnosed with Functional Class I-III Osteoarthritis of the knee or hip
* Patient has required treatment of target joint pain within the 90 days prior to study start and met at least one of the following: was unable to consistently control target joint pain with non-opioid pain reliever, unable to treat target joint pain with non-opioid pain reliever because treatment was contraindicated per investigator judgement, or had received an opioid(single or combination product) for treatment of target joint pain, with the equivalent of less than or equal to 40 mg/day of oral morphine sulfate, inclusive of breakthrough pain medication
* Patient has reported a target joint pain score of at least 5 (11-point Likert Scale) at baseline

Exclusion Criteria:

* Patient for whom hydromorphone was contraindicated because of a documented history of an allergic reaction (hives, rash, etc) or a clinically significant intolerance to hydromorphone or other opioids
* Patient requiring treatment with monoamine oxidase inhibitors, or receiving systemic chemotherapy or had an active malignancy of any type or had clinically significant abnormalities in clinical chemistry, hematology or urinalysis, or had a documented history of gout, pseudogout, Paget's disease, fibromyalgia
* uncontrolled inflammatory arthritis or NSAID-dependent inflammatory arthritis or any chronic pain syndrome that could interfere with the assessment of pain and/or other symptoms of osteoarthritis
* Patient who is pregnant and/or breastfeeding
* Patient with a documented history of drug abuse/dependence/misuse or narcotic analgesic abuse/dependence/misuse, or unable to discontinue all formulations of prior pain medications (opioid and/or non-opioid) during the washout period of the study
* Patient who had a documented history of a medical condition, which, in the investigator's opinion, could compromise the patient's ability to swallow, absorb, metabolize, or excrete study drug, including (but not limited to) intractable nausea and/or vomiting, and/or severe gastrointestinal narrowing

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2003-11; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Time-interval weighted AUC pain ratio (AUC/by an individual's maximum possible benefit AUC)using Baseline Observation Carried Forward imputation(up to Week 12); AUC was the cumulative pain intensity differences from baseline (titration and maintenance).

SECONDARY OUTCOMES:
WOMAC pain subscale for the AUC ratio and change from baseline at each time point; Index score and other subscale analyzed using the AUC ratio and change from baseline (no imputation, BOCF and LOCF imputation); Other included MOS Sleep Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- See also: A Phase 3, Randomized, Double-Blind, Fixed-Dose, Parallel-group Comparison of Controlled-Release Hydromorphone HCl vs. Placebo in Patients with Osteoarthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=123&filename=CR013273_CSR.pdf